CLINICAL TRIAL: NCT03751943
Title: Clinical Investigation of NanoFUSE® Bioactive Matrix and Autogenous Bone in Posterolateral Spinal Fusion (Nonloadbearing)
Brief Title: NanoFUSE® PL Gutter PMCF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NanoFUSE Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR-00001
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Degenerative Disc Disease
Keywords: Demineralized Bone Matrix; Primary Lumbar Fusion; Autograft Lumbar Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- NanoFuse® PL Gutter (Other): NanoFUSE® Bioactive Matrix (75%) w/autograft (25%) within one posterolateral gutter (unilateral)
  Interventions: Device: NanoFUSE® Bioactive Matrix (75%) w/autograft (25%)

INTERVENTIONS:
Device: NanoFUSE® Bioactive Matrix (75%) w/autograft (25%) — NanoFUSE® Bioactive Matrix (75%) w/autograft (25%)within one posterolateral gutter

SUMMARY:
This study is a Post Market Follow Up Study to compare the fusion rates between the NanoFUSE® Bioactive Matrix (75%) w/autograft (25%) and autogenous bone in posterolateral gutter spinal fusion.

DETAILED DESCRIPTION:
NanoFUSE® is indicated to be placed into bony voids or gaps of the skeletal system that are not intrinsic to the stability of the bony structure (i.e. the posterolateral spine and pelvis.) These defects may be surgically created osseous defects created from traumatic injury to the bone. NanoFUSE® must be used with autograft as a bone graft extender in the posterolateral spine. This product provides a bone graft substitute that remodels into the recipient's skeletal system. Radiographic success will be the primary judgement of success. All patient's achieving fused or probably fused status will be judged as a success.

ELIGIBILITY:
Inclusion Criteria:

* Grade I or II (less than 50% slip f the cephalic vertebra compared to the caudal vertebra) degenerative spondylolisthesis at one or two contiguous levels between L1 and L5
* Lumbar spinal stenosis at the same levels of the degenerative spondylolisthesis producing radiculopathy or neurogenic claudication unresponsive to a minimum of 3 months of nonsurgical treatment, or such patients with worsening neurological condition
* Patients who are medically suitable for surgical management and the use of NanoFUSE® Bioactive Matrix is consistent with product labeling
* Patients who have consented for surgical treatment
* Patients able to provide informed consent for the study and complete the questionnaires

Exclusion Criteria:

* Lytic spondylolisthesis
* Non degenerative stenosis (example: tumor, trauma, epidural, lipomatosis)
* Segmental kyphosis at the level of the spondylolisthesis
* Rheumatoid arthritis
* Active infection
* On long term disability or workers compensation claim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Radiographic Success | 12 months
  All patients achieving fused or probably fused status will be judged as successes at 12 months.

SECONDARY OUTCOMES:
Overall patient success | 12 months postoperatively
  Overall patient success will be based on all clinical and radiographic evaluation parameters and complications for the indication for use.
  Success criteria includes the following:
  * Presence of radiographic fusion as evidenced by identification of new bone mass
  * No hardware failure or screw blackout
  * Decreased level of pain (VAS)
  * Maintained or improved level of function (ODI)
  * Maintained or improved neurological status

IPD SHARING:
Plan to Share IPD: Undecided